CLINICAL TRIAL: NCT05312918
Title: Large Scale Transition to a Dolutegravir-based First-line ART in the South: Virological Response and Impact on HIV Drug Resistance in a Real Life Context (DoReaL Study)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: CIRBA, Abidjan, Ivory Coast (Unknown); SEREFO, Bamako, Mali (Unknown); BIOLIM/FSS/UL, Lomé, Togo (Unknown)
Responsible Party: Sponsor
Other Study IDs: ANRS 12427 DoReaL
Record Dates: First submitted 2021-09-22; First posted 2022-04-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: HIV Infections
Keywords: HIV Infections; Dolutegravir; HIV drug resistance; Real Life
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood samples will be collected for this study and will be used for viral load testing and drug resistance evaluation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Main objective The main objective of the study is to assess the virological efficacy of a Dolutegravir-based first-line ART in use under real-life conditions in national programs in resource-limited settings in patients infected with HIV-1 and initially under a NNRTI-based first-line, and determine the impact of NRTI resistance on the success of the new strategy.

Secondary objectives

* Determine the level of virological suppression (HIV-1 RNA <200 copies/ml) at 6, 12 and 24 months after transition from an NNRTI first-line to a DTG first-line.
* Determine the level of virological suppression at the WHO threshold (HIV-1 RNA <1000 copies/ml).
* To determine the frequency of development of resistance and the profiles of mutations in patients with virological failure (HIV-1 RNA ≥200 copies/ml) and the potential impact on the 2nd line strategies combining DTG and currently recommended by the WHO.
* To determine the impact of pre-transition resistance to NRTIs on the virological suppression under DTG first-line and on the development of resistance to integrase inhibitors.
* Study pre-transition resistance acquired under DTG first-lines at the thresholds of 20% and 5% of the viral population, respectively using Sanger and Ultra-deep Sequencing (UDS) approaches.

Identify program factors associated with virological failure and/or the development of drug resistance.

DETAILED DESCRIPTION:
Antiretroviral therapy (ART) has dramatically changed the pronostic of HIV/AIDS infection over the last 20 years, by reducing the mortality and morbibidity associted with the infection. This is mostly true in sub-Saharan African, the most affected region of the world. The UNAIDS 2019 report confirms this fact, and shows a significant reduction in the number of deaths related to HIV infection as access to antiretrovirals (ARV) increases. However, in the absence of cure by current treatments, the management and treatment of the infection should still be considered for life. This makes this management complex and challenging. Indeed, the risk of failure to treatment is real, this risk is accompanied by that of developing resistance to treatment, which should lead to a change in treatment. The limited number of molecules therefore requires the development of strategies that must be effective in maintaining virological suppression for as long as possible and should also limit the emergence and circulation of resistant viruses. To address these priorities, the World Health Organization (WHO) recommends since 2016, the introduction of a first-line ART more efficient and more robust, combining molecules with a high genetic barrier to resistance. In its latest 2019 recommendations for resource-limited countries, WHO recommends a first-line ART comprising two nucleoside reverse transcriptase inhibitors (NRTIs) and one integrase inhibitor (INI), preferably tenofovir (TDF)+Lamivudine (3TC )/emtricitabine (FTC)+dolutegravir (DTG). This new strategy is expected in the context of sub-Saharan Africa, where the increase of pre-treatment and acquired HIV drug resistance has been worrying for several years, but raises a certain number of uncertainties. Indeed, available and published data on the effectiveness of DTG are mainly from studies conducted in Northern countries, very few clinical trials have evaluated or are underway to evaluate the strategy in Southern countries and virtually no evaluation of the effectiveness of this approach in the context of real life in the South has been conducted to date. In addition, few or no recommendations have been made to accompany this transition to a new DTG-based first-line in the South. This is of greater concern for patients who are currently under non-NRTI-based first-line , and who will be switched to a new DTG-based first-line. This population will certainly include very variable virological profiles, ranging from patients in virological suppression, to patients who are not virologically suppressed, with potential accumulation of resistance mutations. In the absence of clear and funded recommendations for the organization of these transitions, the risk of this transition producing results below expectations is real and significant. In addition, the reality of the management of HIV infection in the South regularly faces significant challenges associated with limited financial and human resources. This often makes it difficult to apply decisions made even at the national level. For illustration, despite the unanimity around the use of viral load for monitoring people on ART, access to and the availability of this test in daily practice remains challenging in many countries. It is therefore essential to evaluate the virological response in people who will be switched from the current first-line, to the new first-line, in real life conditions, in the South. This study, developed and considered as a priority by the AC43 working group "Medical Virology" of the ANRS, aims to evaluate this new strategy in real life context in three countries of sub-Saharan Africa, Côte d'Ivoire, Mali and Togo. The main objective is to assess the virological efficacy of the DTG-based first-line in real life conditions, for patients initially receiving an NNRTI-based first-line, followed-up in the national programs and determine the impact of baseline NRTI-drug resistance on the success of the new strategy. All these three countries have adopted the new WHO recommendations and the deployment of the DTG-based first-line is being initiated. It is therefore essential that this research be conducted along side with this ongoing transition, so that the results will help developping adequate recommendations that will allow programs in the South to better organise the transition, to improve the therapeutic and virological monitoring of patients, to prevent early failures, and the emergence and rapid circulation of drug resistance.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or over.
* Infected with HIV-1.
* On an NNRTI-based first-line for at least 6 months.
* Initiating a new 1st line ART based on DTG according to national recommendations.
* Agree to participate in the study and provide free, written and informed consent.

Exclusion Criteria:

* Infection with HIV-2 or HIV1+2.
* Ongoing participation in another virological study on HIV infection

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: HIV-1 infected individuals who are transitioning from an NNRTI-based first-line to a Dolutegravir-based first-line treatment.
Sampling Method: Non-Probability Sample
Enrollment: 603 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Proportion virological success | 48 weeks
  Proportion of patients with virological success at Week 48 (Month 12), defined by a VL <200 copies/ml.

SECONDARY OUTCOMES:
Virological suppression at W24 (VL< 200 copies/ml) | 24 weeks
  Proportion of patients with virological suppression at W24 (VL< 200 copies/ml).
Virological suppression at W96 (VL< 200 copies/ml) | 96 weeks
  Proportion of patients with virological suppression at W96 (VL< 200 copies/ml).
Virological suppression at VL thresholds of 200 copies/ml, considering the first point of viral load and the control viral load if the first point of viral load was >200 copies/ml. | 36 weeks
  Proportion of patients with virological suppression at VL thresholds of 200 copies/ml, considering the first point of viral load at W24 and the control viral load at W36 if the first point of viral load was >200 copies/ml.
Virological suppression at VL thresholds of 200 copies/ml, considering the first point of viral load and the control viral load if the first point of viral load was >200 copies/ml. | 60 weeks
  Proportion of patients with virological suppression at VL thresholds of 200 copies/ml, considering the first point of viral load at W48, and the control viral load at W60 if the first point of viral load was >200 copies/ml.
Virological suppression at VL thresholds of 200 copies/ml, considering the first point of viral load and the control viral load if the first point of viral load was >200 copies/ml. | 108 weeks
  Proportion of patients with virological suppression at VL thresholds of 200 copies/ml, considering the first point of viral load at W96, and the control viral load at W108 if the first point of viral load was >200 copies/ml.
Virological suppression at the WHO threshold (< 1000 copies/ml). | 24 weeks
  Proportion of patients with virological suppression at the WHO threshold at W24 (< 1000 copies/ml).
Virological suppression at the WHO threshold (< 1000 copies/ml). | 48 weeks
  Proportion of patients with virological suppression at the WHO threshold at W48 (< 1000 copies/ml).
Virological suppression at the WHO threshold (< 1000 copies/ml). | 96 weeks
  Proportion of patients with virological suppression at the WHO threshold at W96 (< 1000 copies/ml).
Virological suppression at VL thresholds of 1000 copies/ml, considering the first point of viral load, and the control viral load if the first point of viral load was >1000 copies/ml. | 36 weeks
  Proportion of patients with virological suppression at VL thresholds of 1000 copies/ml, considering the first point of viral load at W24, and the control viral load at W36 if the first point of viral load was >1000 copies/ml.
Virological suppression at VL thresholds of 1000 copies/ml, considering the first point of viral load, and the control viral load if the first point of viral load was >1000 copies/ml. | 60 weeks
  Proportion of patients with virological suppression at VL thresholds of 1000 copies/ml, considering the first point of viral load at W48, and the control viral load at W60 if the first point of viral load was >1000 copies/ml.
Virological suppression at VL thresholds of 1000 copies/ml, considering the first point of viral load, and the control viral load if the first point of viral load was >1000 copies/ml. | 108 weeks
  Proportion of patients with virological suppression at VL thresholds of 1000 copies/ml, considering the first point of viral load at W96, and the control viral load at W108 if the first point of viral load was >1000 copies/ml.
Virological suppression at the optimal threshold (<50 copies/ml) | 24 weeks
  Proportion of patients with virological suppression at the optimal threshold at W24 (<50 copies/ml)
Virological suppression at the optimal threshold (<50 copies/ml) | 48 weeks
  Proportion of patients with virological suppression at the optimal threshold at W48 (<50 copies/ml)
Virological suppression at the optimal threshold (<50 copies/ml) | 96 weeks
  Proportion of patients with virological suppression at the optimal threshold at W96 (<50 copies/ml)
Virological suppression at VL thresholds of 50 copies/ml, considering the first point of viral load, and the control viral load if the first point of viral load was >50 copies/ml. | 36 weeks
  Proportion of patients with virological suppression at VL thresholds of 50 copies/ml, considering the first point of viral load at W24, and the control viral load at W36 if the first point of viral load was >50 copies/ml.
Virological suppression at VL thresholds of 50 copies/ml, considering the first point of viral load, and the control viral load if the first point of viral load was >50 copies/ml. | 60 weeks
  Proportion of patients with virological suppression at VL thresholds of 50 copies/ml, considering the first point of viral load at W48, and the control viral load at W60 if the first point of viral load was >50 copies/ml.
Virological suppression at VL thresholds of 50 copies/ml, considering the first point of viral load, and the control viral load if the first point of viral load was >50 copies/ml. | 108 weeks
  Proportion of patients with virological suppression at VL thresholds of 50 copies/ml, considering the first point of viral load at W96, and the control viral load at W108 if the first point of viral load was >50 copies/ml.
Proportion of patients with virological suppression at VL thresholds of 50, 200 copies/ml and 1000 copies/ml, depending on the viral load at the time of switch | 24 weeks
  Proportion of patients with virological suppression at VL thresholds of 50, 200 copies/ml and 1000 copies/ml, at W24, depending on the viral load at the time of switch according to 3 groups (VL of D0 <200 copies/ml, between 200 and 1000 copies/ml, and ≥1000 copies/ml)
Proportion of patients with virological suppression at VL thresholds of 50, 200 copies/ml and 1000 copies/ml, depending on the viral load at the time of switch | 48 weeks
  Proportion of patients with virological suppression at VL thresholds of 50, 200 copies/ml and 1000 copies/ml, at W48, depending on the viral load at the time of switch according to 3 groups (VL of D0 <200 copies/ml, between 200 and 1000 copies/ml, and ≥1000 copies/ml)
Proportion of patients with virological suppression at VL thresholds of 50, 200 copies/ml and 1000 copies/ml, depending on the viral load at the time of switch | 96 weeks
  Proportion of patients with virological suppression at VL thresholds of 50, 200 copies/ml and 1000 copies/ml, at W96, depending on the viral load at the time of switch according to 3 groups (VL of D0 <200 copies/ml, between 200 and 1000 copies/ml, and ≥1000 copies/ml)
Frequency of drug resistance | 24 weeks
  Frequency of resistance mutations acquired at confirmed virological failure, at VL thresholds of 200 copies/ml and 1000 copies/ml.
Profiles of resistance mutations | 24 weeks
  Profiles of resistance mutations acquired at confirmed virological failure, at VL thresholds of 200 copies/ml and 1000 copies/ml.
Frequency of drug resistance | 48 weeks
  Frequency of resistance mutations acquired at confirmed virological failure, at VL thresholds of 200 copies/ml and 1000 copies/ml.
Profiles of resistance mutations | 48 weeks
  Profiles of resistance mutations acquired at confirmed virological failure, at VL thresholds of 200 copies/ml and 1000 copies/ml.
Frequency of drug resistance | 96 weeks
  Frequency of resistance mutations acquired at confirmed virological failure, at VL thresholds of 200 copies/ml and 1000 copies/ml.
Profiles of resistance mutations | 96 weeks
  Profiles of resistance mutations acquired at confirmed virological failure, at VL thresholds of 200 copies/ml and 1000 copies/ml.
GSS (Genotypic susceptibility score) | 24 weeks
  Proportion of patients with a GSS ≤1 at W24
GSS (Genotypic susceptibility score) | 48 weeks
  Proportion of patients with a GSS ≤1 at W48
GSS (Genotypic susceptibility score) | 96 weeks
  Proportion of patients with a GSS ≤1 at W96.
Frequency of pre-transition resistance mutations to NRTIs | At baseline, before DTG initiation
  Frequency of pre-transition resistance mutations to NRTIs
Proportion of HIV minority variants | Up to 108 weeks.
  Proportion of minority variants (5% threshold) in patients with resistance mutations to NRTIs and/or DTG in the event of virological failure.

CONTACTS AND LOCATIONS:
Overall Officials: Avelin AGHOKENG, Study Director — IRD 224 - CNRS 5290 - UM1-UM2; Anoumou Claver DAGNRA, Study Director — BIOLIM - FSS - UL
Locations (3):
- CIRBA, Abidjan, Côte d’Ivoire
- SEREFO, Bamako, Mali
- Biolim/Fss/Ul, Lomé, Togo